CLINICAL TRIAL: NCT01921049
Title: Systemic Inflammatory Response Syndrome (SIRS) in Patients Undergoing Major Procedures in Oral and Maxillofacial Surgery
Status: Completed | Type: Observational
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Dr. Wolfgang A. Wetsch, M.D., University of Cologne
Other Study IDs: 13-229
Record Dates: First submitted 2013-08-06; First posted 2013-08-13 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2014-12

CONDITIONS: Systemic Inflammatory Response Syndrome (SIRS)
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No

SUMMARY:
Patients undergoing major procedures in oral and maxillofacial surgery more often develop a systemic inflammatory response syndrome (SIRS) in the first days of postoperative critical care therapy than patients with a comparable major surgery in other regions. The reasons for this finding are unknown and have not been studied in depth so far. We hypothesize that surgical trauma in this region might activate pro-inflammatory pathways. By examining the proteome of patients at different stages (prior to the surgery, at ICU admission, on the second postoperative day and when SIRS has ended clinically), we aim to identify the involved pro-inflammatory pathways and identify possible target proteins that might be clues to modification of postoperative SIRS in the future.

ELIGIBILITY:
Inclusion Criteria:

* age 18-99yrs
* scheduled for elective surgery with risk for development of SIRS
* written and informed consent

Exclusion Criteria:

* age <18yrs
* pregnancy
* emergency surgery
* failure to obtain patient consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients undergoing major procedures in oral and maxillofacial surgery during the study period
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2013-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
change of concentration of pro-inflammatory cytokines [µg/l] | up to 10 days post surgery
  Change of concentration of pro-inflammatory cytokines from pre-operative sample over icu-admission, 2nd postoperative day and clinical end of SIRS.

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang A. Wetsch, M.D., Principal Investigator — Department of Anaesthesiology and Critical Care Medicine, University Hospital of Cologne
Locations (1):
- Department of Anaesthesiology and Critical Care Medicine, University Hospital of Cologne, Cologne, Germany